CLINICAL TRIAL: NCT04170842
Title: Music During Paediatric Outpatient Wound Dressing Changes: Impact on Anxiety, Pain and Patient Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: CIRB 2016-2565
Record Dates: First submitted 2019-11-03; First posted 2019-11-20 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-10

CONDITIONS: Wound Heal
Keywords: Wound dressing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music intervention (Experimental): The music intervention used in the study will be a patient selected list of songs or other music delivered to the participant by passive listening via in-ear or on-ear headphones. They will be given the choice of using their own personal headphones or use a pair provided by the hospital. If choosing to use a hospital device, the earphones provided will be disposable to minimise infection risk from re-use.
  Patient preferred music has shown to be more effective than preselected, or prescriptive music. Prescriptive music, if not of the patient's preference, could cause further discomfort, distress or anxiety. Therefore, investigators will use streaming services to provide a bank of music containing a wide range of music and genres to suit the majority of music preferences. Music will also be curated based on feedback from age-appropriate sources to identify common and popular music in the target participant age group.
  Interventions: Other: Music intervention
- Control (No Intervention): Wound dressing procedure conducted according to clinical practice

INTERVENTIONS:
Other: Music intervention — Participants will work with the music therapist to make their selections. Music therapists will provide input on how best to synchronise type, tempo and genre of music to the wound dressing procedure. As musical preference is very personal, the choice of music provided will try to strike a balance of providing what is acceptable to patients while not exposing them to music with known stimulatory effects.
  Arms: Music intervention

SUMMARY:
Background: Wound dressing changes can be painful and distressing for children and the consequences of poorly managed pain and anxiety can be lifelong. Multiple sessions are usually required, and recurrent painful episodes can trigger significant anxiety and behavioural changes with subsequent escalation on re-exposure. Music has been shown to improve relaxation and reduce autonomic activity in paediatric oncology outpatients and have significant positive effect on postoperative pain, anxiety and distress.

Aims: The investigators propose using music listening as a complement to alleviate anxiety, reduce pain and improve the experience of surgical outpatients undergoing wound dressing changes. Investigators will also evaluate the impact on physiological parameters, such as heart rate and blood pressure.

Hypothesis: That pain and anxiety are significantly reduced and patient satisfaction is significantly improved when wound dressings are accompanied by music intervention.

Methodology: A prospective crossover randomised controlled trial recruiting 88 surgical outpatients aged 9 years and above undergoing multiple wound dressing changes. Patients will be randomised to receive music intervention either during the first or subsequent dressing change, with the alternate dressing change not accompanied by music. Patient selected music will be chosen with the input of a trained music therapist. Participants will complete post session self-assessment questionnaires on pain, anxiety and satisfaction. Physiological parameters will be measured pre and post session.

Importance: If proven feasible and effective, this intervention may improve patient experience by reducing pain and anxiety associated with outpatient wound dressing changes, improve patient satisfaction by taking advantage of the relaxing and calming effects of music listening, and improve clinical efficiency by using a cost-effective method for alleviating pain and anxiety

Risks/benefits: There is minimal risk as usual standard treatment protocols for wound management continues. Patients may benefit from the soothing effects of music.

DETAILED DESCRIPTION:
Music intervention - The music intervention used in the study will be a patient selected list of songs or other music delivered to the participant by passive listening via in-ear or on-ear headphones. They will be given the choice of using their own personal headphones or use a pair provided by the hospital. If choosing to use a hospital device, the earphones provided will be disposable to minimise infection risk from re-use.

Patient preferred music has shown to be more effective than preselected, or prescriptive music. Prescriptive music, if not of the patient's preference, could cause further discomfort, distress or anxiety. Therefore, investigators will use streaming services to provide a bank of music containing a wide range of music and genres to suit the majority of music preferences. Music will also be curated based on feedback from age-appropriate sources to identify common and popular music in the target participant age group.

Participants will work with the music therapist to make their selections. Music therapists will provide input on how best to synchronise type, tempo and genre of music to the wound dressing procedure. As musical preference is very personal, the choice of music provided will try to strike a balance of providing what is acceptable to patients while not exposing them to music with known stimulatory effects.

Patients will be given the opportunity to look to music therapists for support in choosing or creating a playlist to accompany their procedure.Through a brief questionnaire the music therapists will gather pertinent information such as favourite styles, experience playing instruments, favourite artists/songs as well as the challenges related to their first experience. The music therapist will help to identify possible song choices/playlists for various parts of the procedure that may decrease their perception of pain by refocusing their attention.

Randomisation - This will be a randomised crossover study. Patients will be randomised into 2 groups:

Group 1: One dressing change or procedure after recruitment will be accompanied by music intervention. Subsequent dressing change or procedure will NOT be accompanied by music intervention.

Group 2: One dressing change or procedure after recruitment will NOT be accompanied by music intervention. Subsequent dressing change or procedure will be accompanied by music intervention.

With this crossover design, all recruited participants will have the opportunity to experience the music intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 9 years and above, male or female
2. Anticipated to require at least 2 further wound dressing changes or outpatient painful procedures (e.g. cryotherapy for skin lesions)
3. Already had at least one outpatient dressing change or painful outpatient procedure prior to recruitment
4. Able to communicate clearly, navigate simple technical software, be awake and alert
5. Not hearing impaired
6. Willing to use headphones
7. Able to read and communicate in English

Exclusion Criteria:

1. Hearing impaired
2. Abnormal anatomy of external ear (unable to use headphones)
3. Wound site prevents use of headphones - for example, on the ear

Ages: 9 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2016-12-23 (Actual); Primary Completion 2019-03-25 (Actual); Study Completion 2019-03-28 (Actual)

PRIMARY OUTCOMES:
Self-assessment of pain | Immediately after intervention
  Using the numeric rating score, which is standard pain score used in the institution ranging from 0-10 where a score of 10 indicates 'worst possible pain' and 0 indicates 'no pain'.
Anxiety score | Immediately after intervention
  Spielberger State-Trait Anxiety Inventory Score for Children (STAIC) which is a validated anxiety score in children, or the Spielberger STAI Score which is a validated anxiety score in adolescents and adults. This score allows adjustment for the different scores that may be produced for a given situation in individuals who may vary in baseline anxiety levels.
Satisfaction survey | Immediately after intervention
  A modified version of the patient satisfaction survey currently used by KK Hospital to assess patient satisfaction with outpatient services

SECONDARY OUTCOMES:
Heart rate | Before and immediately after intervention
  Physiological observations before and after dressing changes
Blood pressure readings | Before and immediately after intervention
  Physiological observations before and after dressing changes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stinson J, Yamada J, Dickson A, Lamba J, Stevens B. Review of systematic reviews on acute procedural pain in children in the hospital setting. Pain Res Manag. 2008 Jan-Feb;13(1):51-7. doi: 10.1155/2008/465891. PMID 18301816
- [Background] Hyland EJ, D'Cruz R, Harvey JG, Moir J, Parkinson C, Holland AJA. An assessment of early Child Life Therapy pain and anxiety management: A prospective randomised controlled trial. Burns. 2015 Dec;41(8):1642-1652. doi: 10.1016/j.burns.2015.05.017. Epub 2015 Oct 6. PMID 26452308
- [Background] Wilson-Smith EM. Procedural Pain Management in Neonates, Infants and Children. Rev Pain. 2011 Sep;5(3):4-12. doi: 10.1177/204946371100500303. PMID 26526331
- [Background] Stouffer JW, Shirk BJ, Polomano RC. Practice guidelines for music interventions with hospitalized pediatric patients. J Pediatr Nurs. 2007 Dec;22(6):448-56. doi: 10.1016/j.pedn.2007.04.011. PMID 18036465
- [Background] George S, Ahmed S, Mammen KJ, John GM. Influence of music on operation theatre staff. J Anaesthesiol Clin Pharmacol. 2011 Jul;27(3):354-7. doi: 10.4103/0970-9185.83681. PMID 21897507
- [Background] Moris DN, Linos D. Music meets surgery: two sides to the art of "healing". Surg Endosc. 2013 Mar;27(3):719-23. doi: 10.1007/s00464-012-2525-8. Epub 2012 Oct 6. PMID 23052506
- [Background] Tan X, Yowler CJ, Super DM, Fratianne RB. The efficacy of music therapy protocols for decreasing pain, anxiety, and muscle tension levels during burn dressing changes: a prospective randomized crossover trial. J Burn Care Res. 2010 Jul-Aug;31(4):590-7. doi: 10.1097/BCR.0b013e3181e4d71b. PMID 20498613
- [Background] Protacio J. Patient-directed music therapy as an adjunct during burn wound care. Crit Care Nurse. 2010 Apr;30(2):74-6. doi: 10.4037/ccn2010250. No abstract available. PMID 20360454
- [Background] van der Heijden MJ, Oliai Araghi S, van Dijk M, Jeekel J, Hunink MG. The Effects of Perioperative Music Interventions in Pediatric Surgery: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. PLoS One. 2015 Aug 6;10(8):e0133608. doi: 10.1371/journal.pone.0133608. eCollection 2015. PMID 26247769
- [Background] DeLoach Walworth D. Procedural-support music therapy in the healthcare setting: a cost-effectiveness analysis. J Pediatr Nurs. 2005 Aug;20(4):276-84. doi: 10.1016/j.pedn.2005.02.016. PMID 16030507